CLINICAL TRIAL: NCT00128232
Title: Safety and Efficacy of Octreotide LAR in Treatment Naïve Acromegalic Patients
Brief Title: Safety and Efficacy of Octreotide Long Acting Release (LAR) in Treatment Naïve Acromegalic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995B2401
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Acromegaly
Keywords: Acromegaly; untreated; newly diagnosed; octreotide LAR
MeSH Terms: conditions — Acromegaly

INTERVENTIONS:
Drug: Octreotide LAR

SUMMARY:
Currently, the first line treatment for acromegaly is surgery, in order to remove the adenoma causing overproduction of growth hormone which leads to acromegaly. Octreotide LAR is approved for treatment of acromegaly after surgery if the disease is not controlled. This study was aimed to test the safety and efficacy of octreotide LAR in acromegalic patients who did not have any previous treatment for acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or previously untreated acromegalic patients
* Lack of suppression of growth hormone (GH) nadir to <1.0 µg/L, after oral administration of 75g of glucose (oral glucose tolerance test [OGTT])
* Insulin-like growth factor-I (IGF-I) levels above the upper limits of normal, i.e. 97th percentile (adjusted for age and gender)

Exclusion Criteria:

* Requires surgery for recent significant deterioration in visual fields or other neurological signs, which are related to the pituitary tumor mass
* No evidence of pituitary adenoma on magnetic resonance imaging (MRI)
* Symptomatic cholelithiasis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-12; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Mean GH and IGF-I at baseline, week 12, 24 and 48

SECONDARY OUTCOMES:
Tumor volume at baseline, week 24 and 48
Signs and symptoms of acromegaly at baseline, week 12, 24 and 48
Safety and tolerability at any time on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Petersenn, MD, Principal Investigator — Universität Duisburg-Essen